CLINICAL TRIAL: NCT06935955
Title: Helicobacter Pylori Gastritis and Its Relation to Metabolic Syndrome Components
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Mohmmed, demonstrator, Assiut University
Other Study IDs: Helicobacter Pylori Gastritis
Record Dates: First submitted 2025-04-07; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Gastritis
MeSH Terms: conditions — Gastritis | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- cohort 1 gastritis patients: The study will include 114 patients diagnosed with gastritis in the Gastroenterology unit and scheduled for upper gastrointestinal endoscopy with stomach biopsy
  Interventions: Diagnostic Test: upper endoscopy

INTERVENTIONS:
Diagnostic Test: upper endoscopy — All subjects will be asked to complete a medical history questionnaire, followed by physical examination (height, body weight, waist circumference and blood pressure), and laboratory investigations (fasting blood glucose, liver function test, total cholesterol, triglycerides, low-density lipoprotein cholesterol and high-density lipoprotein cholesterol( The endoscopy will be carried out by the same specialist, with assessment of chronic and acute gastritis, atrophic gastritis and metaplasia. The endoscopist will obtain five biopsies samples, two from the antrum, two from the corpus and one from incisura.
  All biopsies will be processed at the Pathology Department laboratory and embedded in paraffin blocks. For histological examination, two sets of tissue sections will be stained: one with hematoxylin and eosin (H&E) and the other with Giemsa stain. Each sample will undergo a double-blind review by two independent pathologists according to the USS (HP, neutrophils, mononuclear cells, atro

SUMMARY:
2.2 Aim

1. To evaluate the association between H. pylori infection and the components of metabolic syndrome.
2. To assess the relationship between the histopathologic features of chronic gastritis evaluated using USS and the components of metabolic syndrome in both H. pylori-positive and H. pylori-negative patients.

2.4. 2- Study Setting: Department of Pathology, Faculty of Medicine, Assiut University.

c. Sample Size Calculation: Sample size was calculated using Epi- Info7. Based on The H. pylori-positive patients were more likely to develop dyslipidemia, and 77.47% of individuals testing positive for H. pylori have higher total cholesterol levels (11). With a confidence limit of 5% and a confidence level of 80%, the minimum number of patients required for this study is 114 cases

2.4.4 -Study tools The study will include 114 patients diagnosed with gastritis in the Gastroenterology unit and scheduled for upper gastrointestinal endoscopy with stomach biopsy. Written informed consent will be obtained from all patients participating in the study.

All subjects will be asked to complete a medical history questionnaire, followed by a physical examination (height, body weight, waist circumference, and blood pressure) and laboratory investigations (fasting blood glucose, liver function test, total cholesterol, triglycerides, low-density lipoprotein cholesterol, and high-density lipoprotein cholesterol( The endoscopy will be carried out by the same specialist, and it will assess chronic and acute gastritis, atrophic gastritis, and metaplasia. The endoscopist will obtain five biopsy samples: two from the antrum, two from the corpus, and one from the incisura.

All biopsies will be processed at the Pathology Department laboratory and embedded in paraffin blocks. For histological examination, two tissue sections will be stained: hematoxylin and eosin (H&E) and Giemsa stain. Each sample will undergo a double-blind review by two independent pathologists according to the USS (HP, neutrophils, mononuclear cells, atrophy, and intestinal metaplasia), and each variable will be graded semi-quantitatively.

Statistical analysis using suitable tests will be used to assess our results.

2.4.5 -Research outcome measures:

1. Primary (main): to evaluate the association between H.pylori gastritis and its relation to metabolic syndrome components
2. Secondary (subsidiary):

2.5-Data management and analysis : Data collection All subjects will be asked to complete a medical history questionnaire, followed by a physical examination (height, body weight, waist circumference, and blood pressure) and laboratory investigations (fasting blood glucose, liver function test, total cholesterol, triglycerides, low-density lipoprotein cholesterol, and high-density lipoprotein cholesterol.

Computer software Statistical package for social science (SPSS) program v. 25 (IBM, August 2017).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above with dyspeptic symptoms

Exclusion Criteria:

* People who have a history of H.Pylori eradication or gastric surgery.
* Those who have already received anti-cholesterol therapy.
* Those suffering from severe liver disease, severe kidney disease, or cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 114 patients diagnosed with gastritis in the Gastroenterology unit and scheduled for upper gastrointestinal endoscopy with stomach biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Dyslipidemia | periprocedural
  we will measure Low-density lipoprotein and serum cholesterol as a marker of dyslipidemia